CLINICAL TRIAL: NCT00348543
Title: Prophylactic Laser Treatment of Drusen Maculopathy in Age-related Macular Degeneration.
Brief Title: Prophylactic Laser Treatment of Drusen Maculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 97346
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 1999-10

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macula degeneration; prophylactic laser treatment; exudative complication
MeSH Terms: conditions — Macular Degeneration | interventions — Laser Therapy

INTERVENTIONS:
Procedure: laser treatment

SUMMARY:
To study the effect of mild laser treatment on the incidence of exudative complications in soft drusen maculopathy. We hypothesise that mild laser treatment causing a proliferation of the retinal pigment epithelium and enhancing the capacity of clearing drusen material from Bruch's membrane.

ELIGIBILITY:
Inclusion Criteria:

* > 55 years of age,
* Soft drusen maculopathy,
* VA 0.8-1.0

Exclusion Criteria:

* VA <0.8,
* Pigment clumps,
* PED,
* CNV,
* Atrophy,
* Haemorrhage,
* Diabetes retinopathy,
* Sign cataract,
* Glaucoma

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1999-12; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity

SECONDARY OUTCOMES:
incidence of exudative complications

CONTACTS AND LOCATIONS:
Overall Officials: Christina I Frennesson, MD, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Dept of Ophthalmology, Linköping University, Linköping, Sweden